CLINICAL TRIAL: NCT02147119
Title: Radial Artery Function Following Trans-radial Cardiac Catheterisation
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PG13/32/30205
Record Dates: First submitted 2014-04-07; First posted 2014-05-26 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients post- cardiac catheterisation
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography

SUMMARY:
The investigators will study Radial artery injury and endothelial function following trans-radial cardiac catheterisation. Radial artery injury will be quantified pre- and post- angiography using Optical Coherence Tomography. The participants will also have radial endothelial function assessed using flow-mediated dilatation at baseline, 24 hours, one week, one month and three months post- angiography. Blood will be taken pre and 24 hours post angiography for characterisation of endothelial progenitor cell numbers and function. The hypothesis is that trans-radial catheterisation will cause a reduction in flow-mediated dilatation which peaks at 24 hours and recovers at three months. The investigators hope to correlate the rate of this recovery with peri-procedural progenitor cell numbers.

ELIGIBILITY:
Inclusion Criteria:

* Stable outpatient population aged between 18-85 attending for trans-radial cardiac catheterisation

Exclusion Criteria:

* Recent myocardial infarction (<3 months)
* Severe aortic stenosis
* Chronic renal failure (eGFR<30)
* Inability to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable outpatient population attending for angiography
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Flow-mediated dilatation | baseline, 24 hours, one week, four weeks and three months post-angiography
  Radial artery flow-mediated dilatation will be assessed at the above stated time points

SECONDARY OUTCOMES:
Radial artery injury | Baseline and up to 1 hour Post angiograpy sheath insertion
  Optical coherence tomography examination of the radial artery will be made at baseline and following sheath insertion.
Endothelial progenitor cell number an function Endothelial progenitor cell number and function | Baseline and at 24 hours post-angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Mitchell, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical research facility University Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Derived] Mitchell A, Fujisawa T, Mills NL, Brittan M, Newby DE, Cruden NLM. Endothelial Progenitor Cell Biology and Vascular Recovery Following Transradial Cardiac Catheterization. J Am Heart Assoc. 2017 Oct 28;6(11):e006610. doi: 10.1161/JAHA.117.006610. PMID 29080864